CLINICAL TRIAL: NCT04003545
Title: Application of LED Photobiomodulation in the Treatment of Chronic Low Back Pain: a Randomized, Double-blind Clinical Trial
Brief Title: Application of LED Photobiomodulation in the Treatment of Chronic Low Back Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TFilippo
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In the placebo group, the laser application will be simulated in the same way as the active group, but the device will be turned off.
  The outcome assessor will not know to which group the patients belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): Thirty eight patients will be recruited from UNINOVE outpatient units and randomly allocated in the two groups.
  Interventions: Radiation: LED Photobiomodulation
- Placebo group (Placebo Comparator): Thirty eight patients will be recruited from UNINOVE outpatient units and randomly allocated in the two groups.
  Interventions: Other: Placebo LED Photobiomodulation

INTERVENTIONS:
Radiation: LED Photobiomodulation — A total of twelve laser applications (3 sessions per week) will be provided to the patients as treatment. A LED board with wavelengths of 660nm and 850nm at 5mW of power will be used for 30 minutes, resulting in a total energy of 3J per point in each session. The application site will be the lumbar region, in contact with the skin. The LED cluster (light-emitting diodes) has 72 LEDs.
  Arms: Active group
Other: Placebo LED Photobiomodulation — For the placebo group, the procedures will be the same, however the LED equipment will remain off.
  Arms: Placebo group

SUMMARY:
Lumbar pain, or low back pain, may be defined as pain or discomfort located from the lower portion of the costal margin to the gluteal folds, with or without referred pain in the legs. This pain is classified as non-specific lumbar pain when its cause is unknown, as well as chronic when it persists for longer than three months with the appearance of disabilities for activities of daily life. Treatments for low back pain are usually pharmacological, focusing on analgesics, muscle relaxants and anti-inflammatories. Although protective factors, such as exercise, healthy diet and functional training may mitigate the evolution of pain, physical disability due to pain and functional loss reduce quality of life. Photobiomodulation (PBM) can be defined as the therapeutic use of light sources to reduce inflammation and relief pain. In this context, the objectives of this study are to develop and evaluate the effectiveness of an application protocol of an LED cluster for the treatment of chronic low back pain in a randomized, double-blind clinical trial that will be conducted in the outpatient facility of Universidade Nove de Julho (Uninove). Patients with chronic nonspecific low back pain, who signs the Informed Consent Form approved by the Uninove Institutional Review Board will be included in the study. Treatment sessions will be performed with a LED cluster three times a week for 4 weeks (totaling 12 sessions) in the lumbar region, and the outcomes will be measured with the following evaluations: VAS - Visual Analog Scale; Roland-Morris Disability Questionnaire (RMDQ); Schöber test; Modified Oswestry Disability Questionnaire and Algometry.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of vertebral pain that do not respond to symptomatic treatment with anti-inflammatory drugs for at least 3 months;
* Moderate to severe pain measured by Visual Analogue Scale (VAS> 4);
* Diagnosis of chronic nonspecific low back pain (as previously defined);
* Signed Informed Consent Form to participate in the study and availability to visit the clinic for treatment and evaluations.

Exclusion Criteria:

* Presence of other osteomuscular and rheumatic diseases;
* Presence of symptoms and signs of osteomioarticular disease, even if without known diagnosis;
* Clinical signs and complaints of osteomioarticular pain in the lower limbs (hips and ankles), as well as in spinal region;
* Use of Photobiomodulation up to 90 days before the inclusion;
* Clinical signs of neuropathy, including radiculopathy and peripheral nerve injury;
* Presence of systemic inflammatory diseases (rheumatoid arthritis, Reiter arthritis, spondylitis ankylosing, generalized polyarthritis, neoplasia);
* Presence of metabolic or endocrine diseases;
* Presence of Fibromyalgia;
* Presence of serious psychiatric disorders with demands for specialist care;
* Use of steroids injections up to 48 hours before inclusion;
* Infection or tumor in the area of Photobiomodulation application;
* Presence of severe blood dyscrasias;
* Presence of blood clotting disorders (including local thrombosis);
* Use of oral anticoagulant;
* Presence of Affective Psychotic Disorder that hinders adherence to the treatment;
* History of lumbar surgery;
* Patients who submit to government benefits due to low back pain.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in low back pain assessed by VAS (visual analog scale) | Baseline (Before the first application of LED) and 4 weeks after (after the last application).
  Patients will be present with a 10-cm ruler in which 0 means total absence of pain and 10 the maximum pain.

SECONDARY OUTCOMES:
Change in disability assessed by Roland-Morris Disability Questionnaire (RMDQ) | Baseline (Before the first application of LED) and 4 weeks after (after the last application).
  This scale assesses physical abilities and psychological factors of patients, inquiring about functional changes of people with low back pain. It presents 24 questions about the conditions of the patient that characterize the presented incapacity. In all questions the phrase "because of my back" is added, and when it comes to answering them, the patient signals only the phrases that best suits him or her at that moment, otherwise the patient should go on to the next sentence. The total count of the marked items can range from a minimum of zero, considered no functional impairment, to a maximum of 24, high functional impairment.
Change in range of motion assessed by Schöber test | Baseline (Before the first application of LED) and 4 weeks after (after the last application).
  the patient will remain in the orthostatic position while the examiner positions his thumbs at the lower margin of the posterior superior iliac spine (PSIS) and draws a horizontal line in the midline between these two structures.
  Then, the examiner firmly holds the tip of a measuring tape against the patient's skin on the marked line and marks a second line 15 cm above the first. The patient is then asked to flex the anterior trunk without increasing pain and a new measurement is marked between the lower and upper marks; finally, the patient returns to the neutral position. The difference between the initial distance (between the two marks on the skin in the neutral position) and the new measurement in the flexed position indicates the mobility of the lumbar spine in centimeters, with precision of millimeters.
Change in disability assessed by Modified Oswestry Disability Questionnaire | Baseline (Before the first application of LED) and 4 weeks after (after the last application).
  The Brazilian version of the Oswestry questionnaire allows the evaluation of the functional disability reported by the patients, based on the level of pain during different activities of daily life. This questionnaire contains ten questions about daily activities for evaluating the impact of pain on the performance of such activities. The results range from zero (minimum disability) to 100 (evident disability).
Change in Pressure Pain Threshold | Baseline (Before the first application of LED) and 4 weeks after (after the last application).
  The Pressure Pain Threshold (PPT) will be evaluated with the J Tech algometer (XXX). The algometer is a hand device with a 1cm² diameter rod and a rubber cover in its tip. It allows the recording, through the electronic device, the pressure applied on a surface. For this evaluation, a pressure will be applied at a constant rate of 1kg/sec to the level at which pain or discomfort is reported by the volunteer who will be lying on a stretcher. The evaluated muscles will be: gluteus medius; tensor fasciae latae; tibialis anterior; proximal ischiotibial (ischium); paravertebral muscle (lumbar L2-L5 and sacral S1-S3).